CLINICAL TRIAL: NCT02092155
Title: TGF-B as a Marker of Pleurodesis in Patients With Tunneled Pleural Catheters
Brief Title: Biomarker Levels During Indwelling Pleural cAtheter Sample Testing
Acronym: BLAST
Status: Enrolling by invitation | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00044267
Record Dates: First submitted 2014-03-17; First posted 2014-03-20 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Malignant Pleural Effusions
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pleural fluid attained during drainage of indwelling pleural catheter
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Indwelling tunneled pleural catheter

SUMMARY:
Some patients that have a tunneled pleural catheter will not have the pleural fluid (water around the lung) return after some time (pleurodesis). The purpose of this study is to understand how the investigators can predict who will achieve pleurodesis and how this occurs by studying the pleural effusion.

DETAILED DESCRIPTION:
An alternative and emerging treatment for malignant pleural effusions is the placement of a chronic indwelling pleural catheter.

Tunneled pleural catheters (TPC) are ideal for treatment of malignant pleural effusion (MPE) associated with a trapped or non-expandable lung which will not have sufficient visceral and parietal pleura apposition for chemical pleurodesis. Transforming growth factor-Beta 1 (TGF-β) is a profibrotic cytokine, and a potent inducer of Plasminogen activator inhibitor-1 (PAI-1) in human pleural mesothelial cells. PAI-1 inhibits protease-dependent fibrinolytic activity and along with TGF-β, its concentration is increased in exudative and tuberculous pleural effusion. TGF-β levels in pleural fluid have been shown to correlate with pleural thickness in tuberculosis pleurisy and empyema in rabbits.

TGF-β is a multifunctional cytokine primarily produced by mesothelial cells in the pleural space, but can also originate from lung parenchymal macrophages that migrate to the pleural space. In humans, TGF-β consists of three isoforms (TGF-β1, TGF-β2, and TGF-β3). They share many biological activities and their actions on cells are qualitatively similar in most cases. TGF-β stimulates the extracellular matrix production and studies support that TGF-β over-production is a key regulator in pleural fibrosis and chemical pleurodesis. Moreover, TGF-β signaling for the production of PAI-1 is clearly noted in human mesothelial cells of different origins. Different inflammatory stimuli in the pleural space including malignancy and infection may activate TGF-β up-regulation and enhanced production which in turns results in PAI-1 expression.

ELIGIBILITY:
Inclusion criteria:

* Pleural effusion (etiology fulfilling one of the following criteria):

  1. Malignant effusion confirmed by cytology or pleural biopsy
  2. exudative effusion in the setting of known malignancy with no other identifiable cause
  3. Malignant effusion due to tumors that are historically rapidly responsive to systemic therapy (small cell lung cancer, hematological malignancies) will only be included if refractory to standard chemotherapy
* 18 years of age
* Symptoms such as shortness of breath, cough, or chest fullness/chest discomfort
* Demonstration of symptomatic improvement after therapeutic thoracentesis
* Recurrent pleural effusion after therapeutic thoracentesis
* Capacity to provide informed consent

Exclusion criteria:

* Projected life expectancy less than 30 days.
* Radiographic evidence of trapped lung - persistent lung collapse with failure of the majority (>50%) of the lung to reexpand following drainage of a pleural effusion
* Previous lobectomy or pneumonectomy on the affected side
* Patient receiving intrapleural chemotherapy
* Chylothorax - pleural effusion with triglyceride levels > 110 mg/dl or chylomicrons on lipoprotein analysis, most commonly due to trauma/obstruction of the thoracic duct
* Parapneumonic effusion - pleural effusion associated with pneumonia
* Empyema - infected pleural space as defined by purulent pleural fluid, positive gram stain, or positive culture
* Inability to adequately perform pleural drainage at home
* Uncorrectable bleeding disorder
* Skin infection at the site of intended catheter insertion
* Pregnant women - detected by spot urine testing prior to the procedure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the interventional pulmonology team who receive indwelling pleural catheters for a malignant pleural effusion.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2014-01; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To determine the median time to pleurodesis | 12 week follow up
  Duration of follow-up will be 12 weeks. After 12 weeks, all patients who do not achieve spontaneous pleurodesis will adhere to the standard drainage protocol.

SECONDARY OUTCOMES:
TGF-B levels over time | 12 weeks
  To determine the threshold TGF-B level to determine accuracy of predicting auto-pleurodesis

CONTACTS AND LOCATIONS:
Overall Officials: Lonny Yarmus, DO, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States